CLINICAL TRIAL: NCT06130176
Title: Single-step Functional Sinus Endoscopy and Transoral Surgery Enhance Odontogenic Sinusitis Treatment Outcomes: a Randomized Controlled Trial
Brief Title: Single-step Functional Sinus Endoscopy and Transoral Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qassim University (Other)
Collaborators: Beni-Suef University (Other); Tanta University (Other)
Responsible Party: Principal Investigator, Ghada Amin Khalifa, PhD, Professor of Maxillofacial Surgery and Diagnostic Science, Qassim University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: # REC-FDBSU/02062022-03/EM
Record Dates: First submitted 2023-11-07; First posted 2023-11-14 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2024-08

CONDITIONS: Maxillary Sinusitis
Keywords: Maxillary Sinusitis; Odontogenic Maxillary Sinusitis
MeSH Terms: conditions — Maxillary Sinusitis

STUDY DESIGN:
Intervention Model Description: The OMS will be treated with Single-step Functional Sinus Endoscopy and Transoral Surgery via department-integrated therapy
Who Masked: Participant, Investigator
Masking Description: This study will be double blinded randomized control trail. The patients and investigators who will collect the data will not be informed about the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Single-step Functional Sinus Endoscopy and Transoral Surgery (Experimental): The patients who will be included in this study will be treated by functional sinus endoscopy and transoral surgery to remove the dental cause in the same visit to treat odontogenic sinusitis. The functional sinus endoscopy will be performed by the otolaryngologist, while the transoral surgery will be performed by oral and maxillofacial surgeon.
  Interventions: Procedure: Single-step Functional Sinus Endoscopy and Transoral Surgery
- Functional sinus endoscopy (Active Comparator): The patients who will be included in this study will be treated by functional sinus endoscopy to treat odontogenic sinusitis, and it will be performed by the otolaryngologist.
  Interventions: Procedure: Functional sinus endoscopy
- Trans oral Surgery (Active Comparator): The patients who will be included in this study will be treated by transoral surgery to treat odontogenic sinusitis, and it will be performed by by oral and maxillofacial surgeon
  Interventions: Procedure: Trans oral Surgery

INTERVENTIONS:
Procedure: Single-step Functional Sinus Endoscopy and Transoral Surgery — In each patient, the operation will be carried out by an otorhinolaryngologist and a maxillofacial surgeon. The procedures of the functional sinus endoscopy (FSE) will performed as follow: Under general anesthesia, the origin of the turbinate, and the lateral nasal wall will be conducted. The following stage will be infundibulotomy, which ensures that the uncinate process will be completely removed. The ostium will be dilated with a Stammberger dilatator starting with a 0-degree endoscope then shift to a 30- or 45-degree endoscope to clean the sinus. The cavity will be irrigated after removal of the odontogenic diseases and the purulent discharge will suctioned.In addition to FSE, the maxillofacial surgeon will conduct the necessary oral surgery procedures.The needed transoral procedures will be tooth extraction, oro-antral fistula closure or cystectomy.
  Other Names: FSE/OS
  Arms: Single-step Functional Sinus Endoscopy and Transoral Surgery
Procedure: Functional sinus endoscopy — All patients in this group will only be treated with FSE, which will be conducted by an otolaryngologist. The FSE procedures will be carried out in the same way as the group of Single-step Functional Sinus Endoscopy and Transoral Surgery.
  Other Names: FSE
  Arms: Functional sinus endoscopy
Procedure: Trans oral Surgery — Every patient in this group will only be treated with transoral surgical procedures to remove dental pathology. Oral and maxillofacial surgeons will undertake these treatments. The procedure will be either tooth extraction, oro-antral fistula closure, or cystectomy. If extraction is not needed, endodontic treatment will be performed to remove necrotic pulp. The oro-antral fistula will be closed in two layers using a buccal advanced flap and a palatal rotational flap. In the case of odontogenic cysts, the lesion will be removed by raising a trapezoidal flap.
  Other Names: OS
  Arms: Trans oral Surgery

SUMMARY:
Dento- alveolar or dental structural diseases that affect the floor of the maxillary sinus can cause maxillary sinusitis which is known as odontogenic maxillary sinusitis (OMS). Many treatment protocols have been documented to treat OMS. However, There is no unanimity among clinicians on how and who should treat OMS, whether is it otolaryngologist, oral/maxillofacial surgeons, or dentist. Therefore, this study will be will be enrolled to evaluate the efficacy of the Single-step Functional Sinus endoscopy and trans-oral surgery in the management of maxillary sinusitis raised from Odontogenic origin via Department- integrated therapy.

DETAILED DESCRIPTION:
The OMS is a well-known but understudied kind of sinusitis that necessitates a treatment regimen different from non-odontogenic sinusitis. It requires specialized attention because it differs in its pathophysiology, microbiology, diagnosis, and therapy than other forms of non-odontogenic sinusitis. There are several surgical techniques have been published to treat odontogenic maxillary sinusitis, such as transoral, transnasal endoscopic, or combined techniques. Multiple specialists are daily facing patients with maxillary sinusitis either odontogenic or non-odontogenic, including otolaryngologist, maxillofacial/oral, and dental surgeons.

The direct transoral method, which involves making a bone window in the anterolateral maxillary wall, is more familiar to maxillofacial/oral surgeons, whereas the transnasal endoscopic approach is gaining favor, particularly among otolaryngologists. There is no unanimity among clinicians on how and who should treat OMS, whether it is otolaryngologist, maxillofacial, or oral surgeon. This is one of the reasons why the results are frequently challenged as reported by others. Therefore, this study will be will be enrolled to evaluate the efficacy of the Single-step Functional Sinus endoscopy and trans-oral surgery in the management of maxillary sinusitis raised from Odontogenic origin via Department- integrated therapy.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of OMS that is not responding to dental treatment and/or medical treatment
2. Agreement on the odontogenic cause between an ENT specialist and a dentist/maxillofacial surgeon (There is bone loss surrounding the tooth's root and a connection between the dental lesion and sinus on CT scans)
3. Availability of clinical, radiographic, and ESS data.

Exclusion Criteria:

1. Maxillary sinus malignancy
2. Sinuses with a previous surgery
3. Non-odontogenic Sinusitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2018-11-11 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Thickness of the sinus mucosa | Two weeks after intervention
  On coronal and sagittal CT scans, the thickness of the sinus mucosa will be measures by using measuring tool of the CT scan machine. For each of these picture sets, six mucosal thickness measurements will be taken. Then the average of these measurements will be calculated
Thickness of the sinus mucosa | One month after intervention
  On coronal and sagittal CT scans, the thickness of the sinus mucosa will be measures by using measuring tool of the CT scan machine. For each of these picture sets, six mucosal thickness measurements will be taken. Then the average of these measurements will be calculated
Thickness of the sinus mucosa | Three monthsafter intervention
  On coronal and sagittal CT scans, the thickness of the sinus mucosa will be measures by using measuring tool of the CT scan machine. For each of these picture sets, six mucosal thickness measurements will be taken. Then the average of these measurements will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Ghada A Khalifa, professor, Principal Investigator — College of Dentistry, Qassim University, Saudi Arabia
Locations (1):
- Ghada Amin Khalifa, Buraidah, Qassim Province, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting six months after publication
Access Criteria: IPD will be shared up on request by sending to the corresponding author